CLINICAL TRIAL: NCT04661124
Title: Evaluation of the Heidelberg Engineering SPECTRALIS With Flex Module for In-vivo Imaging in the Supine Position
Status: Completed | Type: Observational
Sponsor: Heidelberg Engineering GmbH (Industry)
Collaborators: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: S-2018-3
Record Dates: First submitted 2020-12-03; First posted 2020-12-10 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Retinal Disease; Healthy Eyes
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Adult Normal Eyes: see Inclusion/Exclusion criteria; imaged with OCT and/or OCTA
  Interventions: Device: SPECTRALIS; Device: SPECTRALIS with Flex Module
- Adult Pathology Eyes: see Inclusion/Exclusion criteria; imaged with OCT and/or OCTA
  Interventions: Device: SPECTRALIS; Device: SPECTRALIS with Flex Module

INTERVENTIONS:
Device: SPECTRALIS — ophthalmic imaging device with head and chinrest
  Other Names: SPECTRALIS HRA+OCT (and variants) with OCT Angiography Module
Device: SPECTRALIS with Flex Module — ophthalmic imaging device on mobile instrumentation stand
  Other Names: SPECTRALIS HRA+OCT (and variants) with Flex Module

SUMMARY:
This is a prospective clinical study conducted at one clinical site in the United States.

DETAILED DESCRIPTION:
The conducted study is an observational study for an imaging device used in the aid of ophthalmology diagnosis.

ELIGIBILITY:
Adult Normal Eyes Population (AN)

Inclusion Criteria for AN Population

1. Age ≥ 22 years
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions.
3. Physically able to be positioned in all required imaging positions (upright at chinrest and supine).
4. Able to fixate.
5. Best corrected visual acuity ≥ 20/40 in both eyes.

Exclusion Criteria for AN Population

1. Eye with ocular media not sufficiently clear to obtain acceptable study-related imaging.
2. Subjects who cannot tolerate the imaging procedures.
3. Clinically significant ocular disease in either eye as determined by an Investigator.
4. Ocular surgical intervention (except for refractive laser surgery or cataract surgery) in either eye.

Adult Posterior Segment Abnormality Eye Population (AD)

Inclusion Criteria for AD Population

1. Age ≥ 22 years
2. Able and willing to undergo the test procedures, sign informed consent, and follow instructions.
3. Physically able to be positioned in all required imaging positions (upright at chinrest and supine).
4. Able to fixate.
5. Eye with a structural and vascular posterior segment abnormality due to ocular disease and/or trauma.

Exclusion Criteria for AD Population

1. Eye with ocular media not sufficiently clear to obtain acceptable study-related imaging.
2. Subjects who cannot tolerate the imaging procedures.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with healthy eyes (AN), and adults with structural and vascular retinal abnormalities (AD)
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2020-12-10 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2024-04-22 (Actual)

PRIMARY OUTCOMES:
The image quality grade of the acquired images as determined by an independent reading center | through study completion, average of 1 day
  OCT, OCTA and IR cSLO - graded Good (2)/Average (1)/Poor (0)
Agreement in identification of abnormalities of the acquired Standard OCT images between the devices | through study completion, average of 1 day
  based on pre-specified abnormalities
Agreement in identification of abnormalities of the acquired OCTA images between the devices | through study completion, average of 1 day
  based on pre-specified abnormalities

SECONDARY OUTCOMES:
Adverse events | through study completion, average of 1 day
  All AEs

CONTACTS AND LOCATIONS:
Overall Officials: Lejla Vajzovic, MD, Principal Investigator — Duke University
Locations (1):
- Duke Eye Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No